CLINICAL TRIAL: NCT06901141
Title: Effect of Different Kinesio Band Applications on Balance, Ankle Function and Leap: A Randomized Controlled Trial
Brief Title: Effect of Different Kinesio Band Applications on Balance, Ankle Function and Jump
Status: Enrolling by invitation | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Demet Sarıyıldız, PhD(c), Principal Investigator, Medipol University
Other Study IDs: MedipolU1
Record Dates: First submitted 2025-03-16; First posted 2025-03-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-03

CONDITIONS: Ankle (Ligaments); Instability (Old Injury)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research is a scientific research and is about "Effect of Different Kinesio Band Applications on Balance, ankle function and jump". Foot and ankle injuries are one of the most common problems among musculoskeletal injuries. Various methods are used to prevent and treat such injuries. In this study, it is aimed to evaluate the effectiveness of these applications by examining the effects of different kinesio band applications on balance, ankle function and jump. Personal information such as name, surname, height, weight will be obtained by asking the participant. The body mass index will be calculated by dividing the size of the size of the size of the length of the height. Different Kinesio band applications will be made to the participants and the effects of these applications will be evaluated. The equilibrium ability of the participants will be evaluated by Modified Star Excursion Balance Test). Foot and ankle functions In the evaluation, a questionnaire of 29 questions will be used. The jump performance will be determined by measuring the horizontal leap distances of the participants. In this study, the participants will be appointed to random groups. This randomness will be provided by using a system called Randomizer.org over the internet. Thus, each participant will be equal to the chances of being included in one of the 3 different band applications. This method allows the study to be conducted impartially and fairly. All evaluations and practices to be made within the scope of this research do not contain an invasive (surgery, needle, etc.) procedure and no risk or discomfort is foreseen for the participants. However, due to kinesio band applications, temporary effects may occur such as sensitivity or allergic reaction in the skin. If such a situation occurs, the tape will be removed immediately and necessary measures will be taken.

ELIGIBILITY:
Inclusion Criteria:

1- Healthy physiotherapy students between the ages of 18-25

Exclusion Criteria:

1. Hip, knee or foot pathology
2. Any neurological impairment
3. A history of lower limb fractures

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy physiotherapy students between the ages of 18-25
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-05-24 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Foot and ankle ability measure (FAAM) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Devrim Tarakcı, Assoc. Dr., Principal Investigator — İstanbul Medipol University
Locations (1):
- İstanbul Beykent University, Istanbul, Büyükçekmece, Turkey (Türkiye)